CLINICAL TRIAL: NCT03428230
Title: Dose-finding Study of Intrathecal Paracetamol Administered Immediately Before Spinal Anaesthesia With Chloroprocaine HCl 1% for Elective Knee Procedures of Short Duration
Brief Title: Intrathecal Paracetamol Before Spinal Anaesthesia With Chloroprocaine HCl 1% for Short Knee Procedures
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sintetica SA (Industry)
Collaborators: Cross Research S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: PAR.3-01-2017; CRO-17-133 (Other: CROSS Research S.A.)
Record Dates: First submitted 2018-01-23; First posted 2018-02-09 (Actual); Results first posted 2021-06-24 (Actual); Last update posted 2021-06-24 (Actual); Status verified 2021-06

CONDITIONS: Pain, Postoperative
MeSH Terms: conditions — Pain, Postoperative | interventions — Acetaminophen; Saline Solution; Solutions; Injections

STUDY DESIGN:
Intervention Model Description: Eligible patients will be randomised into four treatment groups (15 patients/group) to receive either one of the three single doses of Paracetamol 3% (30 mg, 60 mg, 90 mg) or placebo solution (1 mL, 2 mL, 3 mL) according to the randomised, parallel-group design.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study will be double-blind. Neither the Investigator/co-investigators/study nurses involved in the clinical study procedures, nor will the patients be aware of the administered treatment. At the site, syringes for injection will then be prepared by a person not involved in any other study-related activities where a bias is possible.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30 mg Paracetamol 3% (1 mL) (Experimental): 30 mg Paracetamol 3% (1 mL), solution for injection, single dose by intrathecal injection (IT)
  Interventions: Drug: 30 mg Paracetamol 3% (1 mL); Drug: NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection
- 60 mg Paracetamol 3% (2 mL) (Experimental): 60 mg Paracetamol 3% (2 mL), solution for injection, single dose by intrathecal injection (IT)
  Interventions: Drug: 60 mg Paracetamol 3% (2 mL); Drug: NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection
- 90 mg Paracetamol 3% (3 mL) (Experimental): 90 mg Paracetamol 3% (3 mL), solution for injection, single dose by intrathecal injection (IT)
  Interventions: Drug: 90 mg Paracetamol 3% (3 mL); Drug: NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection
- Placebo, 0.9% saline solution (Placebo Comparator): Placebo, 0.9% saline solution (1 mL, 2 mL or 3 mL), solution for injection, single dose by intrathecal injection (IT)
  Interventions: Drug: Placebo, 0.9% saline solution; Drug: NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection

INTERVENTIONS:
Drug: 30 mg Paracetamol 3% (1 mL) — Single administration by intrathecal injection just before spinal anaesthesia. The injection will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  Arms: 30 mg Paracetamol 3% (1 mL)
Drug: 60 mg Paracetamol 3% (2 mL) — Single administration by intrathecal injection just before spinal anaesthesia. The injections will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  Arms: 60 mg Paracetamol 3% (2 mL)
Drug: 90 mg Paracetamol 3% (3 mL) — Single administration by intrathecal injection just before spinal anaesthesia. The injections will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  Arms: 90 mg Paracetamol 3% (3 mL)
Drug: Placebo, 0.9% saline solution — Single administration by intrathecal injection just before spinal anaesthesia. The injections will be performed according to the hospital procedures. For the intrathecal injection of Placebo followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Placebo will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  Other Names: physiological solution
  Arms: Placebo, 0.9% saline solution
Drug: NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection — Immediately after intrathecal administration of the Paracetamol dose or Placebo, all patients will receive a single intrathecal dose of Chloroprocaine HCl 1% according to the Summary of Product Characteristics indications. Time interval between the 2 administrations should not exceed 2 min.
  Other Names: Ampres 1%

SUMMARY:
This is a phase II, single centre, randomised, parallel-group, double-blind, three doses, placebo-controlled, exploratory efficacy and safety study. The objective of this study is to investigate the efficacy and safety of a single intrathecal injection of Paracetamol 3% (30 mg/mL) administered at 3 doses to 3 active treatment groups, as compared to placebo, for post-operative analgesia in knee procedures up to 40 min duration performed under spinal anaesthesia with Chloroprocaine HCl 1%.

DETAILED DESCRIPTION:
Eligible patients undergoing elective short-duration knee procedures up to 40 min duration will be randomised into 4 treatment groups (15 patients per group) to receive either one of the 3 single doses of Paracetamol 3% (D1: 30 mg, D2: 60 mg, D3: 90 mg) or the placebo solution (P: 0.9% saline solution) by intrathecal injection (IT), according to the randomised, parallel-group design.

Immediately after IT paracetamol or placebo administration, all patients will receive a single IT dose of Chloroprocaine HCl 1% (Non-investigational medicinal product, NIMP) according to the Summary of Product Characteristics indications. The time interval between paracetamol IT and chloroprocaine IT injections should not exceed 2 min.

The study will include a screening phase (Visit 1, Day -21/-1), a treatment phase (IMP IT administration, anaesthesia and surgical procedure: Visit 2, Day 1) and a follow-up phase including an observation period (Visit 3), a final visit and two follow-ups (24 h post-dose and day 7±1).

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent: signed written informed consent before inclusion in the study
2. Sex, age and surgery: male/female patients, 18-80 years old (inclusive), scheduled for short duration (up to 40 min) knee procedures
3. Body Mass Index (BMI): 18 - 32 kg/m2 inclusive
4. ASA physical status: I-III
5. Full comprehension: ability to comprehend the full nature and purpose of the study, including possible risks and side effects; ability to co-operate with the investigator and to comply with the requirements of the entire study.

Exclusion Criteria:

1. Physical findings: clinically significant abnormal physical findings which could interfere with the objectives of the study. Contraindications to spinal anaesthesia. History of neuromuscular diseases to the lower extremities
2. ASA physical status: IV-V
3. Further anaesthesia: patients expected to require further anaesthesia
4. Allergy: ascertained or presumptive hypersensitivity to the active principles (paracetamol and/or ester type anaesthetics) and/or formulations' ingredients or related drugs, non-steroidal anti-inflammatory drugs and/or opioid derivatives; history of anaphylaxis to drugs or allergic reactions in general, which the investigator considers could affect the outcome of the study
5. Chronic pain syndromes: patients with chronic pain syndromes taking opioids, anticonvulsant agents or chronic analgesic therapy
6. Pain assessment: patients anticipated to be unable to make a reliable self-report of pain intensity
7. Diseases: significant history of renal, hepatic, gastrointestinal, cardiovascular, respiratory, skin, haematological, endocrine or neurological diseases that may interfere with the aim of the study; ascertained psychiatric and neurological diseases, sepsis, blood coagulation disorders, severe cardiopulmonary disease, thyroid disease, diabetes, other neuropathies, history or evidence of heart failure. History of severe head trauma that required hospitalisation, intracranial surgery or stroke within the previous 30 days, or any history of intracerebral arteriovenous malformation, cerebral aneurism or CNS mass lesion
8. Medications: medication known to interfere with the extent of spinal blocks for 2 weeks before the start of the study. Paracetamol formulations, other than the investigational product, for 2 weeks before the start of the study and during the study. Hormonal contraceptives for females are allowed. Anti-hypotensive, anti-bradycardia (e.g. ephedrine, atropine, Ringer's solution), anti-haemetic and anti-nausea medications will be allowed
9. Investigative drug studies: participation in the evaluation of any investigational product for 3 months before this study. The 3-month interval is calculated as the time between the first calendar day of the month that follows the last visit of the previous study and the first day of the present study
10. Drug, alcohol: history of drug or alcohol abuse according to the Investigator's opinion
11. Pregnancy and lactation: positive pregnancy test at screening (if applicable), pregnant or lactating women [The pregnancy test will be performed to all fertile women and to all women up to 55 years old, if not in proven menopause (available laboratory test confirming menopause or surgically sterilised)]

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-10-22 (Actual); Study Completion 2019-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Claudio Camponovo, MD, Principal Investigator — Department of Anaesthesiology, Clinica Ars Medica, Via Cantonale, CH-6929 Gravesano, Switzerland
Locations (1):
- Department of Anaesthesiology, Clinica Ars Medica, Gravesano, Switzerland

RESULTS

PARTICIPANT FLOW:
Groups:
- 30 mg Paracetamol 3% (1 mL): 30 mg Paracetamol 3% (1 mL), solution for injection, single dose by intrathecal injection (IT)
  30 mg Paracetamol 3% (1 mL): Single administration by intrathecal injection just before spinal anaesthesia.
  The injection will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection: Immediately after intrathecal administration of the Paracetamol dose or Placebo, all patients will receive a single intrathecal dose of Chloroprocaine HCl 1% according to the Summary of Product Characteristics indications. Time interval between the 2 administrations should not exceed 2 min.
- 60 mg Paracetamol 3% (2 mL): 60 mg Paracetamol 3% (2 mL), solution for injection, single dose by intrathecal injection (IT)
  60 mg Paracetamol 3% (2 mL): Single administration by intrathecal injection just before spinal anaesthesia.
  The injections will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection: Immediately after intrathecal administration of the Paracetamol dose or Placebo, all patients will receive a single intrathecal dose of Chloroprocaine HCl 1% according to the Summary of Product Characteristics indications. Time interval between the 2 administrations should not exceed 2 min.
- 90 mg Paracetamol 3% (3 mL): 90 mg Paracetamol 3% (3 mL), solution for injection, single dose by intrathecal injection (IT)
  90 mg Paracetamol 3% (3 mL): Single administration by intrathecal injection just before spinal anaesthesia.
  The injections will be performed according to the hospital procedures. For the intrathecal injection of Paracetamol followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Paracetamol will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection: Immediately after intrathecal administration of the Paracetamol dose or Placebo, all patients will receive a single intrathecal dose of Chloroprocaine HCl 1% according to the Summary of Product Characteristics indications. Time interval between the 2 administrations should not exceed 2 min.
- Placebo, 0.9% Saline Solution: Placebo, 0.9% saline solution (1 mL, 2 mL or 3 mL), solution for injection, single dose by intrathecal injection (IT)
  Placebo, 0.9% saline solution: Single administration by intrathecal injection just before spinal anaesthesia.
  The injections will be performed according to the hospital procedures. For the intrathecal injection of Placebo followed by the intrathecal injection of the anaesthetic, two needles will be used: one introducer needle, which will serve to introduce the second needle through the skin, plus one intrathecal Pencil point needle (27-G or 25-Gauge or Reganesth or Nizell needle) to which the first syringe containing Placebo will be attached first, followed by the second syringe with the anaesthetic. In this way only one intrathecal puncture will be performed. Lumbar puncture will be done according to the standard hospital procedures.
  NIMP: Chloroprocaine HCl 1% (10 mg/mL), solution for injection: Immediately after intrathecal administration of the Paracetamol dose or Placebo, all patients will receive a single intrathecal dose of Chloroprocaine HCl 1% according to the Summary of Product Characteristics indications. Time interval between the 2 administrations should not exceed 2 min.
Period: Overall Study
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Started | 15 | 15 | 15 | 15
Completed | 15 | 15 | 15 | 15
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution | Total
Number analyzed (Participants) | 15 | 15 | 15 | 15 | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.1 (10.9) | 39.7 (15.5) | 40.1 (12.8) | 45.5 (13.6) | 42.85 (13.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 2 | 2 | 8
  Male | 13 | 13 | 13 | 13 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 15 | 15 | 15 | 15 | 60
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Switzerland | 15 | 15 | 15 | 15 | 15

OUTCOME MEASURES:

1. Primary Outcome: Pain Intensity at Rest Evaluated Using a 0-100 mm VAS
Description: The study primary efficacy measures will be the VAS scores at each predefined time-point after the anaesthetic intrathecal injection until eligibility for home discharge ( VAS scale is 0-100 mm, where 0 is no pain and 100 is maximum pain)
Time Frame: Pain intensity at rest evaluated using a 0-100 mm VAS at baseline (within 30 min before NIMP IT injection, 0 h), 1, 1.25, 1.5, 1.75, 2 h after NIMP IT injection, then every 30 min after NIMP IT injection until eligibility for home discharge.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale
  baseline | 9.6 (20) | 16.9 (17.4) | 18.4 (26.4) | 8.1 (14.8)
  1 hour after NIMP | 0.1 (0.3) | 0.1 (0.5) | 3.4 (11.5) | 0 (0)
  1.25 hour after NIMP | 4.6 (11.4) | 1.9 (5.1) | 6.2 (13.7) | 0.6 (1.3)
  1.50 hour after NIMP | 5.9 (13.2) | 4.5 (10.2) | 16.4 (23.6) | 1.2 (2.1)
  1.75 hour after NIMP | 9.5 (16.5) | 15.1 (16.3) | 21.4 (24.3) | 3.6 (6.1)
  2 hours after NIMP | 14.1 (24.6) | 17.8 (19) | 22.8 (23.2) | 3.9 (8.7)
  2.5 hours after NIMP | 16.9 (22.8) | 8.7 (7.1) | 14.7 (15.8) | 7.2 (8.2)
  3 hours after NIMP | 21 (27.7) | 9.6 (12.8) | 7.3 (13) | 10.4 (15.4)
  3.5 hours after NIMP | 19.7 (21.4) | 6.8 (11.4) | 14.2 (25.7) | 11.4 (16.8)
  4 hours after NIMP | 6.8 (8.3) | 13.3 (18.1) | 15.3 (19.1) | 0 (0)
  4.5 hours after NIMP | 2.5 (3.5) | 0 (0) | 2 (2.6) | 0 (0)
  before discharge | 3.7 (4.7) | 4.1 (5.6) | 2.9 (4.5) | 11.3 (7.7)

2. Secondary Outcome: Pain at Rest AUCt1-t2
Description: AUC t1-t2 is defined as the area under the pain intensity curve at the specified time-intervals
Time Frame: Up to 4 hours after injection
Measure: Mean (Standard Deviation); unit: score on a scale*h
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale*h
  AUC 0-2 hours | 13 (13) | 14.8 (12.5) | 26.4 (30.1) | 4.4 (7.1)
  AUC 0-4 hours | 34.6 (29.6) | 26 (10.9) | 92.2 (69.4) | 49.7 (21.7)

3. Secondary Outcome: Pain at Rest AUClast
Description: AUClast is defined as the area under the pain intensity curve from 0 h up to the last assessment time
Time Frame: Up to 24 hours after injection
Measure: Mean (Standard Deviation); unit: score on a scale*h
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
score on a scale*h | 34 (41.3) | 24.7 (15.7) | 42 (50.3) | 15.7 (23.3)

4. Secondary Outcome: Time to First Postoperative Analgesia (Level 1 or 2)
Description: Postoperatively, patients will be administered an analgesic as needed. Post-operative analgesia could include Ketorolac i.v. [Toradol] 30 mg (level 1 analgesia) and/or Tramadol i.v. 1 mg/kg (level 2 analgesia).
  The administered analgesic (level 1 or 2), analgesic dose and intake frequency will be decided according to the reported surgery-related pain intensity.
  Post-operatively, patients were administered an analgesic, as needed. Post-operative analgesia could include Ketorolac i.v. [Toradol] 30 mg (level 1 analgesia) and/or Tramadol i.v. 1 mg/kg (level 2 analgesia).
Time Frame: Up to 24 hours after surgery
Population: Nine (9) patients in D1, 10 in D2, 8 in D3 and 14 in P treatment group did not require postoperative analgesia and were censored in the time to first post-operative analgesia analysis
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 11 | 8 | 14 | 1
Participants
  0-2 hours | 5 | 3 | 7 | 0
  0-4 hours | 6 | 5 | 7 | 1

5. Secondary Outcome: Partecipants to Received Level 1 Analgesia
Description: Partecipants to received Ketorolac i.v. [Toradol] 30 mg administration (level 1 analgesia)
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 5 | 7 | 1

6. Secondary Outcome: Partecipants Received Level 2 Analgesia
Description: Partecipants received Tramadol i.v. 1 mg/kg administration (level 2 analgesia)
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 2 | 0 | 4 | 0

7. Secondary Outcome: Total Number of Partecipants Receiving Analgesic 1
Description: Total number of partecipants receiving Ketorolac i.v. [Toradol] 30 mg
Time Frame: From surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 5 | 7 | 1

8. Secondary Outcome: Total Number of Partecipants Receiving Analgesic 2
Description: Total Number of Partecipants Receiving Tramadol i.v. 1 mg/kg
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 2 | 0 | 4 | 0

9. Secondary Outcome: Percentage of Patients Requiring Analgesia in the First 2 h After Surgery End
Description: Percentage of patients requiring analgesia (level 1 or level 2) in the first 2 h after surgery end
Time Frame: Form surgery day to 2 hours after surgery end
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 5 | 3 | 7 | 0

10. Secondary Outcome: Percentage of Patients Requiring Analgesia in the First 4 h After Surgery End
Description: Percentage of patients requiring analgesia (level 1 or level 2) in the first 4 h after surgery end
Time Frame: from surgery day to 4 hours after surgery end
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 5 | 7 | 1

11. Secondary Outcome: Percentage of Patients Requiring Analgesia From Surgery End Until Eligibility for Discharge
Description: Percentage of patients requiring analgesia (level 1 or level 2) from surgery end until eligibility for home discharge
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 14
Participants | 6 | 5 | 7 | 1

12. Secondary Outcome: Percentage of Patients Requiring Level 1 Analgesia From Surgery End Until Eligibility for Discharge
Description: Percentage of patients requiring level 1 analgesia from surgery end until eligibility for home discharge
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 6 | 5 | 7 | 1

13. Secondary Outcome: Percentage of Patients Requiring Level 2 Analgesia From Surgery End Until Eligibility for Discharge
Description: Percentage of Patients Requiring Level 2 Analgesia From Surgery End Until Eligibility for Home Discharge
Time Frame: from surgery day to 24 hours after surgery
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 2 | 0 | 4 | 0

14. Secondary Outcome: Percentage of Patients Requiring Supplementary Analgesia, Other Than the Planned Level 1 or 2 Analgesia
Description: Percentage of patients requiring supplementary analgesia, other than the planned level 1 or 2 analgesia
Time Frame: from surgery day to 24 hours after surgery
Measure: Number; unit: participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
participants
  level 1 | 6 | 5 | 7 | 1
  level 2 | 2 | 0 | 4 | 0

15. Secondary Outcome: Percentage of Patients Requiring Rescue Anaesthesia
Description: Percentage of patients requiring rescue anaesthesia
Time Frame: from surgery day to 1 hour after injection
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 14 | 15 | 15 | 14

16. Secondary Outcome: Time to Onset of Spinal Block (i.e. Time to Readiness for Surgery)
Description: Spinal block/Readiness for surgery is defined as the presence of an adequate motor block (Bromage's score ≥ 2) and loss of Pinprick sensation, according to the Investigator's opinion. Time to readiness for surgery is defined as the time from the spinal injection (time 0 h) to achievement of readiness for surgery.
Time Frame: Up to 20 minutes after injection
Measure: Median (Inter-Quartile Range); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 5 [2 to 5] | 5 [3 to 5] | 2 [1 to 5] | 5 [2 to 5]

17. Secondary Outcome: Maximum Sensory Block
Description: Maximum level of sensory block
Time Frame: Intraoperative
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants
  T1 | 0 | 0 | 0 | 0
  T2 | 1 | 0 | 0 | 0
  T3 | 0 | 0 | 0 | 0
  T4 | 0 | 0 | 1 | 1
  T5 | 0 | 1 | 1 | 1
  T6 | 1 | 1 | 1 | 1
  T7 | 0 | 1 | 0 | 0
  T8 | 7 | 0 | 6 | 6
  T9 | 0 | 3 | 2 | 0
  T10 | 3 | 5 | 1 | 4
  T11 | 2 | 3 | 2 | 1
  T12 | 0 | 1 | 0 | 1
  L1 | 1 | 0 | 1 | 0
  L2 | 0 | 0 | 0 | 0
  L3 | 0 | 0 | 0 | 0
  L4 | 0 | 0 | 0 | 0
  L5 | 0 | 0 | 0 | 0
  S1 | 0 | 0 | 0 | 0
  S2 | 0 | 0 | 0 | 0
  S3 | 0 | 0 | 0 | 0
  S4 | 0 | 0 | 0 | 0
  S5 | 0 | 0 | 0 | 0

18. Secondary Outcome: Time to Sensory Block
Description: Time to maximum level of sensory block (bilateral Pinprick test using a 20-G hypodermic needle)
Time Frame: Intraoperative
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 10 [10 to 12] | 10 [8 to 14] | 10 [5 to 10] | 10 [6 to 15]

19. Secondary Outcome: Time to Regression of Spinal Block
Description: Time period from spinal injection to the complete regression of sensory block to S1.
Time Frame: Up to 4 hours after injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 100 [85 to 112] | 100 [78 to 125] | 90 [76 to 95] | 95 [89 to 115]

20. Secondary Outcome: Time to Ambulation
Description: Time to unassisted ambulation
Time Frame: Up to 24 hours after injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 139 [120 to 180] | 115 [65 to 150] | 125 [95 to 170] | 125 [120 to 165]

21. Secondary Outcome: Time to First Urine
Description: Time to first spontaneous urine voiding
Time Frame: Up to 24 hours after injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 155 [122 to 220] | 140 [87 to 205] | 145 [100 to 177] | 150 [125 to 170]

22. Secondary Outcome: Time to Eligibility for Discharge
Description: Time to eligibility for home discharge
Time Frame: Up to 24 hours after injection
Measure: Median (95% Confidence Interval); unit: minutes
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
minutes | 170 [145 to 230] | 165 [132 to 195] | 170 [135 to 200] | 168 [145 to 190]

23. Other Pre Specified Outcome: Number of Participants With Neurological Complications Including TNS
Description: Number of Participants with Neurological Complications Including TNS at 24 h post-dose and at day 7±1
Time Frame: From anaesthetic intrathecal injection up to day 7±1 (i.e. 6±1 days after analgesic/anaesthetic IT injection and surgery)
Measure: Count of Participants; unit: Participants
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
Number analyzed (Participants) | 15 | 15 | 15 | 15
Participants | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events throughout the study 48 hours
Arm/Group | 30 mg Paracetamol 3% (1 mL) | 60 mg Paracetamol 3% (2 mL) | 90 mg Paracetamol 3% (3 mL) | Placebo, 0.9% Saline Solution
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 3/15 | 0/15 | 4/15 | 3/15
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 30 mg Paracetamol 3% (1 mL) (N=15) | 60 mg Paracetamol 3% (2 mL) (N=15) | 90 mg Paracetamol 3% (3 mL) (N=15) | Placebo, 0.9% Saline Solution (N=15)
headache (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 1 (1)
hypotension (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
bradycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-10-16): https://cdn.clinicaltrials.gov/large-docs/30/NCT03428230/Prot_SAP_000.pdf